CLINICAL TRIAL: NCT06999889
Title: Comparative Evaluation Of Periodontal Parameters And Periodontal Status In Individuals Of Different Age Groups With And Without Trauma From Occlusion: A Cross Sectional Study
Brief Title: Comparative Evaluation of Periodontal Status and Periodontal Parameters in Different Age Group Individuals With and Without Trauma From Occlusion.
Status: Not yet recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Ashish kumar perio
Record Dates: First submitted 2025-05-15; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Trauma From Occlusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Test Group-1.: Patients showing positive fremitus test in Age Group-26-35Yrs.
  Interventions: Diagnostic Test: Recording of Periodontal Parameters.
- Test Group-2.: Patients showing positive fremitus test in Age Group-36-45Yrs.
  Interventions: Diagnostic Test: Recording of Periodontal Parameters.
- Control Group-1: Patients showing negative fremitus test in Age Group-26-35Yrs.
  Interventions: Diagnostic Test: Recording of Periodontal Parameters.
- Contrl Group-2: Patients showing negative fremitus test in Age Group-36-45Yrs.
  Interventions: Diagnostic Test: Recording of Periodontal Parameters.

INTERVENTIONS:
Diagnostic Test: Recording of Periodontal Parameters. — Periodontal Parameters recording in terms of various indices,measurements and radiographs.

SUMMARY:
Trauma from occlusion (TFO) is defined as an injury resulting in tissue changes within the attachment apparatus as a result of occlusal forces (Glossary of Periodontic Terms American Academy of Periodontology, 2001) This clinical condition is frequently associated with jiggling forces and results in progressive tooth mobility.Experiments performed in animals like the beagle dog showed some periodontal tissue reactions to increasing tooth mobility. Such as (i) Increase in the width of the periodontal ligament area (ii)Increase in the vascularity,vascular permeability and the migration of leukocytes from the vascular plexus and (iii) the increase in number of osteoclasts lining the marginal alveolar bone of the zone of co destruction . Also, the teeth showing increasing mobility exhibit an enhanced rate of periodontal tissue destruction when exposed to experimentally induced periodontitis When trauma from occlusion is the result of alterations in occlusal forces, it is called as primary trauma from occlusion. When it results from the reduced ability of the Periodontal tissues to resist the occlusal forces ,it is known as secondary trauma from occlusion.One of the clinical sign of TFO include presence of Fremitus which means functional tooth mobility.Aggravation of plaque- related inflammatory periodontal disease by trauma from occlusion is still under question.It is unclear whether TFO occurs primarily in periodontitis patients, or bone loss due to periodontitis leads to TFO in later stages. Review of Literature has further revealed that there is no study conducted on anterior teeth with Fremitus and its relation with periodontal parameters.So, it may be hypothesized that TFO may have impact on Periodontal tissue in different age groups as periodontitis is chronic in nature and time of initiation of the disease could not be identified.Periodontitis is chronic in nature and time of initiation of the disease could not be identified. Recently age dependent distribution of periodontitis was studied and findings reported mean clinical attachment loss increased linearly with age and recession contributed increasingly to CAL with age specially after 45-49years.Therefore reduced periodontium in later stages it may lead to TFO, as compared to early stages of life

DETAILED DESCRIPTION:
Trauma from occlusion (TFO) is defined as an injury resulting in tissue changes within the attachment apparatus as a result of occlusal forces (Glossary of Periodontic TermsAmerican Academy of Periodontology, 2001) This clinical condition is frequently associated with jiggling forces and results in progressive tooth mobility.Experiments performed in animals like the beagle dog showed some periodontal tissue reactions to increasing tooth mobility. Such as (i) Increase in the width of the periodontal ligament area (ii)Increase in the vascularity,vascular permeability and the migration of leukocytes from the vascular plexus and (iii) the increase in number of osteoclasts lining the marginal alveolar bone of the zone of codestruction . Also, the teeth showing increasing mobility exhibit an enhanced rate of periodontal tissue destruction when exposed to experimentally induced periodontitis When trauma from occlusion is the result of alterations in occlusal forces, it is called as primary trauma from occlusion. When it results from the reduced ability of the Periodontal tissues to resist the occlusal forces ,it is known as secondary trauma from occlusion.One of the clinical sign of TFO include presence of Fremitus which means functional tooth mobility. A tooth with fremitus has excess contact, possibly related to a premature contact during habitual centric closure and excursive mandibular movements.The role of trauma from occlusion in periodontal disease relies on the belief that excessive occlusal forces do not initiate destructive chronic periodontitis .Though these forces are capable of causing periodontal injury and To establish relation between trauma from occlusion and periodontitis both should be present in destructive stages otherwise combined lesion can't be reproduced.Primary trauma from occlusion without periodontal inflammation results in no loss of attachment, with preservation of a bone matrix that is able to regenerate in the absence of traumatogenic forces. However, when periodontal inflammation is superimposed with trauma from occlusion, alterations in alveolar bone height and volume are not reverted by elimination of traumatogenic forces, with persistence of clinical mobility and gingival inflammation .Aggravation of plaque- related inflammatory periodontal disease by trauma from occlusion is still under question, and further investigations are necessary to elucidate such an association.It is unclear whether TFO occurs primarily in periodontitis patients, or bone loss due to periodontitis leads to TFO in later stages. Review of Literature has further revealed that there is no study conducted on anterior teeth with Fremitus and its relation with periodontal parameters.

So, it may be hypothesized that TFO may have impact on Periodontal tissue in different age groups as periodontitis is chronic in nature and time of initiation of the disease could not be identified. Recently age dependent distribution of periodontitis was studied and findings reported mean clinical attachment loss increased linearly with age and recession contributed increasinginly to CAL with age specially after 45-49years.Therefore reduced periodontium in later stages it may lead to TFO, as compared to early stages of life

ELIGIBILITY:
Inclusion Criteria:1. Systemically healthy individuals will be screened for TFO including Fremitus, Adaptability to TFO, Mobility, Pathological Migration and Tongue thrusting. 2. Systemically healthy individuals will be enrolled in to Two groups, Test group and Control group of 26-35 and 36-45 age group.

* presence of ≥24 natural teeth

Exclusion Criteria:• Current smokers and Former smokers

* Any systemic disease which influence the periodontal tissue such as diabetes mellitus.
* Systemic condition such as Pregnancy and Lactation.
* Systemic Medication for the past 6 months.
* Patients undergoing orthodontic treatment or treated cases.
* Any missing anterior either maxillary or Mandibular teeth.
* History of systemic antibiotics within last 3 months
* Periapical pathology in anterior teeth.
* Any periodontal treatment within 6 months prior to study
* Any developmental anomaly of anterior teeth.
* Presence of prosthesis in Anterior teeth (Crown and Implant)
* No vertical stops due to missing posterior teeth.
* Patients with tongue thrusting habit.
* Patients with parafunction like Bruxism and Clenching Identified through Interview and occlusal examination.
* Patient with Oral Habits like Biting or Holding Objects between the Teeth.
* Patient having any craniomandibular dysfunction or undergone any treatment for temporomandibular joint.

Ages: 26 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Systemically Healthy Individuals in Age Group 26-35 Yrs and 36-45Yrs.
Sampling Method: Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment level (CAL) ) | average 1 year
  Measured in mm from CEJ
Probing Pocket Depth (PPD) | average 1 year
  Measured in mm from free Gingival margin.
Interproximal Alveolar Bone level(From CEJ) | average 1 year
  Measured from CEJ
Pattern of bone Loss. | average 1 year
  Measured from CEJ

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Kumar, BDS, Principal Investigator — Post Graduate Institute of Dental Sciences ,Rohtak
Locations (1):
- Department of Periodontology ,Post Graduate Institute Of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No